CLINICAL TRIAL: NCT03523949
Title: A Study of the Effectiveness of Pain Neuroscience Education in the Elderly.
Brief Title: Pain Neuroscience Education in Old Adults.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Marc Terradas Monllor, Principal Investigator, University of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: END65
Record Dates: First submitted 2018-04-30; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Pain Neuroscience Education; Elderly; Pain Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PNE. (Experimental): Procedure: This educational intervention is based in the latest evidence of pain neuroscience education, used in multiple rehabilitation programs. Its aim is to change the subject's pain understanding, teaching them the biological processes underneath the pain construct, as a mechanism to reduce itself and its related maladaptive thoughts and behaviors.
  Interventions: Behavioral: PNE

INTERVENTIONS:
Behavioral: PNE — The PNE will be delivered by a physiotherapist in a single, group-based session.

SUMMARY:
The primary objectives of this study are to:

* Evaluate the ability of the older adults to understand the biological processes underneath a pain experience.
* Evaluate their ability to modify their behaviors and beliefs about pain and health.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectivity of a single, group-based session of pain neuroscience education (PNE) on old adults. Participants will be 65 years or older, and they will be recruited from primary care medical clinics, public lectures, community centers and through the word of mouth. The intervention consist in one educational session of pain neuroscience education delivered by a physiotherapist. The study design is a single arm, crossover clinical trial, participants will be assessed in 3 different times (1 month before PNE ,pre-PNE, post-PNE) for knowledge of pain neuroscience, pain attitudes, pain catastrophizing and pain-related fear of movement.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 65 years old or more.
* Able to speak and read in Spanish.

Exclusion Criteria:

* Cognitive impairment. Global Deterioration Scale and Functional Assessment Staging (GDS-FAST) will be used for the screening, excluding the subjects with a level 3 or above in the GDS-FAST scale.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge of Pain Neuroscience. Changes from baseline to immediately after PNE. | baseline, pre-PNE, immediately after PNE
  Participants will be asked to complete the Neurophysiology of Pain Questionnaire (NPQ) (Spanish version)

SECONDARY OUTCOMES:
Pain Attitudes. | baseline, pre-PNE, immediately after PNE
  Participants will be asked to complete the Survey of Pain Attitudes Brief Version (SOPA-B) (Spanish version).
Pain Catastrophism. | baseline, pre-PNE, immediately after PNE
  Participants will be asked to complete the Pain Catastrophizing Scale (PCS) (Spanish version).
Pain-related Fear of Movement. | baseline, pre-PNE, immediately after PNE
  Participants will be asked to complete the Tampa Scale of Kinesiophobia (TSK-11) (Spanish version).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Louw A, Podalak J, Zimney K, Schmidt S, Puentedura EJ. Can pain beliefs change in middle school students? A study of the effectiveness of pain neuroscience education. Physiother Theory Pract. 2018 Jul;34(7):542-550. doi: 10.1080/09593985.2017.1423142. Epub 2018 Jan 8. PMID 29308954
- [Background] Moseley L. Unraveling the barriers to reconceptualization of the problem in chronic pain: the actual and perceived ability of patients and health professionals to understand the neurophysiology. J Pain. 2003 May;4(4):184-9. doi: 10.1016/s1526-5900(03)00488-7. PMID 14622702
- [Background] Cox T, Louw A, Puentedura EJ. An abbreviated therapeutic neuroscience education session improves pain knowledge in first-year physical therapy students but does not change attitudes or beliefs. J Man Manip Ther. 2017 Feb;25(1):11-21. doi: 10.1080/10669817.2015.1122308. Epub 2016 Feb 10. PMID 28855788
- [Background] Louw A, Diener I, Landers MR, Puentedura EJ. Preoperative pain neuroscience education for lumbar radiculopathy: a multicenter randomized controlled trial with 1-year follow-up. Spine (Phila Pa 1976). 2014 Aug 15;39(18):1449-57. doi: 10.1097/BRS.0000000000000444. PMID 24875964
- [Background] Louw A, Butler DS, Diener I, Puentedura EJ. Development of a preoperative neuroscience educational program for patients with lumbar radiculopathy. Am J Phys Med Rehabil. 2013 May;92(5):446-52. doi: 10.1097/PHM.0b013e3182876aa4. PMID 23478459
- [Background] Maguire N, Chesterton P, Ryan C. The Effect of Pain Neuroscience Education on Sports Therapy and Rehabilitation Students' Knowledge, Attitudes, and Clinical Recommendations Toward Athletes With Chronic Pain. J Sport Rehabil. 2019 Jul 1;28(5):438-443. doi: 10.1123/jsr.2017-0212. Epub 2018 Oct 15. PMID 29405811
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Lluch E, Duenas L, Falla D, Baert I, Meeus M, Sanchez-Frutos J, Nijs J. Preoperative Pain Neuroscience Education Combined With Knee Joint Mobilization for Knee Osteoarthritis: A Randomized Controlled Trial. Clin J Pain. 2018 Jan;34(1):44-52. doi: 10.1097/AJP.0000000000000511. PMID 28514231
- [Background] Louw A PT, PhD, Zimney K PT, DPT, Reed J PT, DPT, Landers M PT, DPT, PhD, Puentedura EJ PT, DPT, PhD. Immediate preoperative outcomes of pain neuroscience education for patients undergoing total knee arthroplasty: A case series. Physiother Theory Pract. 2019 Jun;35(6):543-553. doi: 10.1080/09593985.2018.1455120. Epub 2018 Mar 28. PMID 29589782
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Background] Andias R, Neto M, Silva AG. The effects of pain neuroscience education and exercise on pain, muscle endurance, catastrophizing and anxiety in adolescents with chronic idiopathic neck pain: a school-based pilot, randomized and controlled study. Physiother Theory Pract. 2018 Sep;34(9):682-691. doi: 10.1080/09593985.2018.1423590. Epub 2018 Jan 10. PMID 29319386
- [Background] Rufa A PT, DPT, OCS, Beissner K PT, PhD, Dolphin M PT, DPT, MS, OCS. The use of pain neuroscience education in older adults with chronic back and/or lower extremity pain. Physiother Theory Pract. 2019 Jul;35(7):603-613. doi: 10.1080/09593985.2018.1456586. Epub 2018 Mar 30. PMID 29601227